CLINICAL TRIAL: NCT00487721
Title: A Pilot Biomarker Study of Oral Silybin-Phytosome Followed by Prostatectomy in Patients With Localized Prostate Cancer
Brief Title: The Effect of High-dose Silybin-phytosome in Men With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 05-1076.cc
Record Dates: First submitted 2007-06-16; First posted 2007-06-19 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Silymarin; Silybin; milk-thistle extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silibin-Phytosome (Experimental): Subjects in this group will take Silibin-Phytosome 13 grams daily, in three divided doses for 2-10 weeks.
  Interventions: Drug: Silibin-Phytosome
- Control (No Intervention): Patients in this arm will not take any intervention.

INTERVENTIONS:
Drug: Silibin-Phytosome — Subjects will take Silibin-Phytosome for 2-10 weeks. The dose of Silibin-Phytosome is 13 grams daily, in three divided doses. Patients will be asked to mix 1 level teaspoon and 1 heaping ¼ teaspoon of Silybin-Phytosome powder into 6 tablespoons of applesauce for each dose.
  Other Names: Silymarin, silibinin, milk thistle
  Arms: Silibin-Phytosome

SUMMARY:
Silibinin has demonstrated anti-cancer activity in the laboratory for several different cancer types, including prostate cancer. Silibinin was originally obtained from milk thistle. Silybin-Phytosome, an oral form of silibinin, has been tested previously in prostate cancer patients to determine the safety of high-dose treatment. This study is for men with prostate cancer who are planning to have their prostate surgically removed. Participants will be given Silybin-Phytosome three times a day from enrollment in the study until the time of their surgery. Participation in this study will not affect the timing of surgery. We obtain blood and urine samples at the start and completion of the trial in addition to prostate tissue from the surgery. These samples will be analyzed for the effect of Silybin-Phytosome at the end of the study.

DETAILED DESCRIPTION:
Prostate cancer is the most common invasive malignancy and the second leading cause of cancer death in American males. In 2005, an estimated 230,000 men will be diagnosed and 30,000 will die from prostate cancer. The current estimated risk of developing prostate cancer is 1 in 6 men. Carcinogenesis and neoplastic progression of prostate cancer depend on both genetic and epigenetic factors; a multi-step process leads to progression from an androgen-dependent, non-metastatic phenotype to a more malignant, metastatic, androgen-independent phenotype.

Treatment options for localized prostate cancer include watchful waiting, surgical prostatectomy, or targeted irradiation. The latter two treatments can cure cancers that are confined to the prostate gland, yet many patients have occult metastasis at the time of presentation, particularly to the bone or regional lymph nodes.

Advanced prostate cancer with metastases presents a difficult therapeutic problem. Those who have disease progression with hormonal therapy have limited options. Patients initially treated with the combination of a Luteinizing Hormone Releasing Hormone (LHRH) analog and a synthetic antiandrogen occasionally respond to withdrawal of the anti-androgen. Chemotherapy is also an option in this setting, with docetaxel-based therapy having a small survival advantage in patients with hormone refractory prostate cancer.

There is clearly a need for more effective regimens for patients with prostate cancer. With the current limitation in treatment options, there has been a renewed public and scientific interest in the use of less toxic herbal preparations in the treatment of cancer. Herbal supplements may play an especially important role in prostate cancer, considering its high incidence and oftentimes slow progression. However, before physicians can confidently recommend dietary supplementation, further scientific investigation is required.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign an Institutional Review Board (IRB) approved informed consent
2. Age greater than 18 years old
3. Male patients with histologically documented adenocarcinoma of the prostate
4. Life expectancy greater than three months
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
6. Adequate organ function including a total Bilirubin less than or equal to 1.5 mg/dl
7. Planned prostatectomy as treatment for prostate cancer.
8. No known metastatic disease

Exclusion Criteria:

1. Prior definitive treatment for prostate cancer with surgery or radiation therapy
2. Use of an investigational medication or device within one month of initiating study therapy.
3. Prior systemic chemotherapy for prostate cancer or any hormonal therapy for prostate cancer.
4. Any use of hormonal therapy (i.e. luteinizing hormone-releasing hormone analog) or anti-androgen therapy.
5. Any condition or any medication which may interfere with the conduct of the study as determined by the principal investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-08; Primary Completion 2007-09 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Michael Glode, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Background] Flaig TW, Gustafson DL, Su LJ, Zirrolli JA, Crighton F, Harrison GS, Pierson AS, Agarwal R, Glode LM. A phase I and pharmacokinetic study of silybin-phytosome in prostate cancer patients. Invest New Drugs. 2007 Apr;25(2):139-46. doi: 10.1007/s10637-006-9019-2. Epub 2006 Nov 1. PMID 17077998
- [Derived] Flaig TW, Glode M, Gustafson D, van Bokhoven A, Tao Y, Wilson S, Su LJ, Li Y, Harrison G, Agarwal R, Crawford ED, Lucia MS, Pollak M. A study of high-dose oral silybin-phytosome followed by prostatectomy in patients with localized prostate cancer. Prostate. 2010 Jun 1;70(8):848-55. doi: 10.1002/pros.21118. PMID 20127732
- See also: Genitourinary care team at the University of Colorado — http://www.uch.edu/conditions/cancer/urologic-cancer/medical-team/index.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve patients were recruited from the urologic oncology clinic at the University of Colorado Hospital between October of 2006 and October of 2007.
Pre-assignment Details: All patients were newly diagnosed with prostate cancer and planning to pursue surgical radical prostatectomy. Patients were excluded from participation if they had received previous treatment for prostate cancer or if their surgery was scheduled within 14 days.
Groups:
- Silibin-Phytosome: Subjects in this group received silybin-phytosome for 2-10 weeks, depending on the time from enrollment until the time of the prostatectomy. The dose of silybin-phytosome was 13 g daily in three divided doses.
- Control: Subjects in the control arm did not receive any treatment or placebo.
Period: Overall Study
Arm/Group | Silibin-Phytosome | Control
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Since this was a pilot study, the number of patients was selected based on the feasibility of accrual and support, rather than statistical calculations. The results of this study will be considered in the planning of future trials with silibinin.
Groups:
- Total: Total of all reporting groups
Arm/Group | Silibin-Phytosome | Control | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: Years] | 56.5 [46 to 66] | 57.5 [49 to 65] | 57 [46 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Measurable Silibinin Tissue Levels
Description: To determine if measurable silibinin tissue levels are detectable in the prostate glands of men treated with Silybin-Phytosome administered according to the protocol. Analysis of silibinin in human fluid and tissue samples was carried out by Liquid chromatography - mass spectrometric (LC/MS/MS) following liquid extraction. Briefly, sample was extracted in acidified ethyl acetate by vortex. Following centrifugation, the organic layer was evaporated to dryness in a rotary evaporator and the samples were dissolved in acetonitrile/ammonium acetate with acetic acid for analysis. Sample analysis was done using an Applied Biosystems 3200 Q-Trap 1 triple quadrupole mass spectrometer with an Agilent 1100 Liquid Chromatography system and HTC-PAL Leap Autosampler. Quantitation of silibinin in samples was done by internal standard reference and batch analysis verified by the inclusion of spiked quality control samples in the appropriate matrix.
Time Frame: At the time of surgery
Population: Per protocol analysis was used and 6 participants that were enrolled in the study were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Silibin-Phytosome
Number analyzed (Participants) | 6
Participants | 3

ADVERSE EVENTS:
Time Frame: Adverse events were assessed within 7 days of the end of of the study.
Arm/Group | Silibin-Phytosome | Control
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Silibin-Phytosome (N=6) | Control (N=6)
Hospitalization or Prolonged Hospitalization (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Silibin-Phytosome (N=6) | Control (N=6)
Diarrhea (Gastrointestinal disorders) | 3 | 0
Hyperbilirubinemia (Investigations) | 1 | 0

LIMITATIONS AND CAVEATS:
Some end of study blood samples were not obtained due to the timing of surgery, tissue was successfully obtained in all participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes